CLINICAL TRIAL: NCT04552821
Title: Study of Biomarkers in Blood and Alveolar Lavage Fluid Samples of Sepsis Patients Complicated With Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Study of Biomarkers in Patients of Sepsis Complicated With Acute Respiratory Distress Syndrome (ARDS)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tianjin Nankai Hospital (Other)
Responsible Party: Principal Investigator, Jianbo Yu, Department of Anesthesiology, Director, Chief physician, Professor, Doctoral tutor, Tianjin Nankai Hospital
Other Study IDs: NKYY_YXKT_IRB_2020_053_01
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Sepsis; Acute Respiratory Distress Syndrome
Keywords: sepsis; Acute Respiratory Distress Syndrome; metabonomics; biomarkers; oxidative stress; Inflammation
MeSH Terms: conditions — Sepsis; Respiratory Distress Syndrome; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples and alveolar lavage fluid were collected from eligible patients within 24 hours after admission to ICU. The blood samples were collected and then placed in a layer at 4°C and centrifuged at 3000×g for 10 minutes. Then the sample were transferred to a cleaning tube and stored in a -80°C refrigerator, waiting for analysis of oxidation and inflammatory indicators.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Non-sepsis and non-ARDS adults receiving mechanical ventilation
- Sepsis complicated with mild ARDS: Patients who meet the criteria of sepsis-3, and also meet the criteria of Berlin diagnostic for mild ARDS
- Sepsis complicated with moderate/severe ARDS: Patients who meet the criteria of sepsis-3, and also meet the criteria of Berlin diagnostic for moderate/severe ARDS

SUMMARY:
1. Title: Study of Biomarkers in Blood and Alveolar Lavage Fluid Samples of Sepsis Patients Complicated With Acute Respiratory Distress Syndrome (ARDS)
2. Research center: Single-center study.
3. Design of the research: A prospective and cohort study.
4. Object of the research: Patients（age≥18 years）those who meet the diagnostic criteria of sepsis complicated with ARDS and grouped into ARDS group and non-ARDS adults receiving mechanical ventilation as control.
5. Sample size of the research: Not less than 30 patients in each group.
6. Research approach: After admission to ICU, patients who meet the criteria are divided into mild group and moderate/severe group according to the severity of ARDS. In addition, blood and alveolar lavage fluid were collected within 24 hours for metabonomics analysis, and differential metabolites were screened out to prove the differentiation ability of differential metabolites between mild and moderate/severe ARDS patients. Then, MSEA and STITCH analysis were performed, and the relationship between different metabolites, HO-1 protein, oxidative stress and inflammatory markers in serum and alveolar lavage fluid were determined. And whether differential metabolites are associated with 28-day mortality in patients with moderate/severe ARDS.
7. Aim of the research: The metabolomics techniques were used to compare the differences between sepsis patients with mild ARDS and moderate/severe ARDS. And determine the relationship between different metabolites, HO-1 protein, oxidative stress and inflammatory markers, as well as the predictive effect of metabolites on 28-day mortality in patients.
8. Statistical analysis: Analytical study.
9. The estimated duration of the study：1-2 years.

DETAILED DESCRIPTION:
This study is a single-center, prospective, retrospective study. In this study, the serum samples and alveolar lavage fluid of patients with sepsis complicated with ARDS were studied by using high performance liquid chromatography (HPLC) tandem electrospray four-stage rod time-of-flight mass spectrometry (LC-ESI-Q-TOF-MS). Aim to screen out the different metabolites between patients with mild and moderate/severe sepsis complicated with ARDS. HO-1 protein, oxidative stress and inflammatory markers in serum and alveolar lavage fluid were measured simultaneously to explore the relationship between HO-1, oxidative inflammatory markers and metabolic markers. In addition, a biomarker model was established to provide an important reference for assisting ARDS disease management and predicting the adverse outcome of patients with sepsis complicated with ARDS.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Patients with sepsis who meet the criteria for sepsis -3
* Patients complicated with Acute Respiratory Distress Syndrome who meet the Berlin diagnostic criteria
* Agree to participate in this study and sign informed consent

Exclusion Criteria:

* Refuse to participate in this study
* Patient with HIV infection, patients in pregnancy or breast stage
* Patient had chronic respiratory ailments
* Patients are now being included in another study
* In the opinion of the attending physician or researcher, there are other conditions that are not appropriate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult patients with sepsis complicated with ARDS
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2024-06-02 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Multivariate data analysis of the metabolites | an average of 1 year
  Record the different metabolites between the control group and ARDS patients
Multivariate data analysis of the metabolites | 12 months
  Record the different metabolites between the patient with mild ARDS and with moderate/severe ARDS

SECONDARY OUTCOMES:
Screening of differentially expressed metabolites as potential mortality predictors for sepsis complicated with ARDS | an average of 1 year
  Investigated the metabolites to distinguish the non-survivors from the survivors of sepsis complicated with ARDS
Pathway Analysis of the differential metabolites | 12 months
  Screened the differential metabolism pathway between mild ARDS and with moderate/severe ARDS, and screened the differential metabolism pathway between non-survivors and survivors

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Yu, MD,PhD, Study Chair — Tianjin Nankai Hospital
Locations (1):
- Tianjin NanKai hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
All of the individual participant data collected during the trial,after deidentification will be shared.And anyone who wishes to acess the date will be available for any purpose.

REFERENCES:
- [Background] Xu J, Pan T, Qi X, Tan R, Wang X, Liu Z, Tao Z, Qu H, Zhang Y, Chen H, Wang Y, Zhang J, Wang J, Liu J. Increased mortality of acute respiratory distress syndrome was associated with high levels of plasma phenylalanine. Respir Res. 2020 Apr 30;21(1):99. doi: 10.1186/s12931-020-01364-6. PMID 32354336
- [Background] Lin S, Yue X, Wu H, Han TL, Zhu J, Wang C, Lei M, Zhang M, Liu Q, Xu F. Explore potential plasma biomarkers of acute respiratory distress syndrome (ARDS) using GC-MS metabolomics analysis. Clin Biochem. 2019 Apr;66:49-56. doi: 10.1016/j.clinbiochem.2019.02.009. Epub 2019 Feb 16. PMID 30779905
- [Background] Metwaly SM, Winston BW. Systems Biology ARDS Research with a Focus on Metabolomics. Metabolites. 2020 May 19;10(5):207. doi: 10.3390/metabo10050207. PMID 32438561
- [Result] Stringer KA, Serkova NJ, Karnovsky A, Guire K, Paine R 3rd, Standiford TJ. Metabolic consequences of sepsis-induced acute lung injury revealed by plasma (1)H-nuclear magnetic resonance quantitative metabolomics and computational analysis. Am J Physiol Lung Cell Mol Physiol. 2011 Jan;300(1):L4-L11. doi: 10.1152/ajplung.00231.2010. Epub 2010 Oct 1. PMID 20889676
- [Result] Evans CR, Karnovsky A, Kovach MA, Standiford TJ, Burant CF, Stringer KA. Untargeted LC-MS metabolomics of bronchoalveolar lavage fluid differentiates acute respiratory distress syndrome from health. J Proteome Res. 2014 Feb 7;13(2):640-9. doi: 10.1021/pr4007624. Epub 2013 Dec 9. PMID 24289193